CLINICAL TRIAL: NCT03259386
Title: Using Arrays of Microelectrodes Implanted in Residual Peripheral Nerves to Provide Dexterous Control of, and Modulated Sensory Feedback From, a Hand Prosthesis
Brief Title: Movement and Sensation for Advanced Prosthetic Hands
Status: Terminated | Type: Observational
Why Stopped: Problem with obtaining microarrays, which are essential components needed to conduct this study.
Sponsor: Mayo Clinic (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Arizona State University (Other)
Responsible Party: Principal Investigator, Shelley S. Noland, Principal Investigator, Mayo Clinic
Other Study IDs: 14-007456; W81XWH-13-PRORP-TRA (Other Grant/Funding Number: CDRMP)
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Amputation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Transradial or Transhumeral amputees: High-count microelectrode arrays are implanted into the upper limb peripheral nerves of transradial or transhumeral amputees.
  Interventions: Device: Microelectrode array

INTERVENTIONS:
Device: Microelectrode array — Microelectrode array implanted in area of amputation of either transradial or transhumeral amputees. This device is not designed to collect data on safety and effectiveness but rather, the device is a tool to assist in the sensory and motor properties of peripheral nerve stump fibers in amputees and is considered basic physiological research. This study was determined to be IDE exempt by the FDA; the study is considered basic physiological research.

SUMMARY:
The purpose of this study is to learn more information about nerves. This study is also designed to learn how the information in nerves could be used to develop new prosthetic devices.

DETAILED DESCRIPTION:
The general design of the study is broken down into two parts: the pre- and post-implantation schedules:

During the 30 days before implantation the participant will be asked to take home a small computer with an Oculus Rift headset and Leap Motion hand tracker. The participant will be asked to use these items five (5) times a week for 30 minutes a session and interact with a displayed virtual reality environment. In this environment the participant will move their intact hand and the Leap Motion will display the hand movements in the virtual environment with the intact hand movements being mirrored between two hand facsimile. The participant will be instructed to move and stretch both their phantom and intact hand in a mirrored fashion. The purpose of these exercises are to allow the participant to become accustomed to the virtual reality setup (equipment and display) as well as providing a mirror box like effect where the virtual hand facsimile for their phantom hand is mapped to their body.

The second phase of the general design continues for 30-90 days post-implantation. We shall perform electrophysiological recordings from a single microelectrode array implanted into either the median, radial, or ulnar nerve. Neural signals (single and compound action potentials) evoked by variegated movements of the fingers and thumb will be recorded on the implanted microelectrode array. By recording electrical signals from the nerves the investigators hope to decode finger movements in real-time using machine learning algorithms. The participants will be asked to complete tasks in controlled virtual environment during the training phase. The virtual environment, which includes virtual arms and hands, will be presented to the participant via the Oculus rift, a pair of virtual reality goggles. The task will require recording the position of arms in space which will be accomplished using the Vicon motion capture system that will use infra-red reflecting markers attached to the participant's arms. The investigators will also use a marker-less motion capture system, Leap Motion, to track the specific movements of the intact hand. Post training, the investigators aim to perform real-time decoding of finger movements in the virtual reality environments.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has previously undergone a transradial (below elbow) or transhumeral (above elbow) amputation.

Exclusion Criteria:

1. Pregnancy
2. Incarceration
3. Inability to consent
4. Serious, untreated comorbidity
5. Patient is diagnosed with a medical condition(s) that seriously increase the risk of electrode implantation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: These are patients that have previously undergone a transradial or transhumeral amputation.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

PRIMARY OUTCOMES:
Number of subjects for whom the investigators can decode finger movements | From 44-104 days post-implantation
  High-count microelectrode arrays are implanted into upper limb peripheral nerves of transradial and transhumeral amputees. Direct micro-stimulation of peripheral nerves will be done using the microelectrode array.

CONTACTS AND LOCATIONS:
Overall Officials: Shelley Noland, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Phoenix, Arizona
  - Arizona State University, Tempe, Arizona